CLINICAL TRIAL: NCT02739919
Title: Bacterial Analysis of Kidney Stones Removed by Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dirk Lange, Assistant Professor, University of British Columbia
Other Study IDs: H16-00637
Record Dates: First submitted 2016-03-16; First posted 2016-04-15 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2016-11

CONDITIONS: Urolithiasis
Keywords: Kidney stones; Renal Calculi
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified and study coded kidney stone and urine samples are collected, processed and analysed in the research laboratory.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this research is to use a controlled laboratory setting to determine whether bacteria isolated from kidney stones of patients play a role in the formation of non-infectious kidney stones. It is well known that struvite stones are associated with active bacterial infection, however the role of bacteria in the formation of non-infection stones (like calcium oxalate) is not well characterized and there are theories that bacteria are involved in the making of these stones.

DETAILED DESCRIPTION:
Kidney stone disease is common, affecting nearly 10% of the population with increasing prevalence and increasing cost associated to treat this disease. While struvite stones (composed of magnesium, ammonium and phosphate crystals) have been associated with the presence of infection, the association between bacteria and non-infection stones is not well characterized. Previous studies have found bacteria present in stones of patients without active infection and with negative pre-operative urine tests.

There are various compositions of kidney stones, including calcium oxalate, calcium phosphate, struvite and uric acid, with calcium oxalate being the most common. It is well known that struvite stones are associated with active infection, however the role of bacteria in the formation of other types of kidney stones, including calcium oxalate, is not well understood. The investigators hypothesize that bacteria present in the urinary tract of patients without active infection have the ability to facilitate calcium oxalate crystal formation by providing a surface for stones to grow. An understanding of the role of bacteria in the formation of non-infection stones could help prevent stone formation by altering the bacteria present within patients to decrease or eliminate their risk of kidney stone disease.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Diagnosed with or have a high index of suspicion of having a kidney stone and scheduled to undergo percutaneous nephrolithotomy.
* Medically fit for definitive surgical management of stone

Exclusion Criteria:

* Those with medical comorbidities preventing them from safely undergoing definitive surgical therapy.
* Patients who are unable to provide informed consent.
* 18 years old or younger
* Diagnosed with an infection stone
* Urinary tract infection within 3 months before date of operation
* Antibiotic use within 3 month before date of operation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Vancouver General Hospital that are diagnosed with a kidney stone and scheduled to undergo percutaneous nephrolithotomy.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Amount of stone formation in artificial urine with isolated bacteria from non-infection kidney stones compared to control measured using FTIR-Microscopy and SEM (concentration measured in mg/mL). | Through study completion, approximately 2 years
  Bacteria will be isolated from non-infection kidney stones allowed to form a biofilm. Next, the bacteria will be incubated in supersaturated artificial urine to precipitate stone formation in vitro and compared to control urine consisting of the same artificial urine without bacteria. Over time, crystallization in the biofilm will be measured using FTIR-Microscopy and SEM.
Bacteria isolated from non-infection kidney stone compared to those identified on pre-operative urine test quantified by simple serial dilution and CFU counting (measured in CFU/mL) and identified using DNA sequencing. | Through study completion, approximately 2 years
  Bacteria will be quantified using simple serial dilution and CFU counting and identified using DNA sequencing. Bacteria will then be correlated with the bacteria identified on pre-operative urine test.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Lange, MSc, PhD, Principal Investigator — University of British Columbia; Ben H Chew, MD, Study Director — University of British Columbia
Locations (1):
- The Stone Centre, VGH/UBC, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No